CLINICAL TRIAL: NCT02067117
Title: Demonstrate the Lot-to-lot Consistency of 3 Consecutive Batches and to Evaluate the Efficacy and Safety of GC FLU®Pre-filled Syringe Injection and 'GC FLU®Injection' Administration.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GCFLU_P4
Record Dates: First submitted 2014-01-19; First posted 2014-02-20 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Prevention of Influenza
Keywords: influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- influenza split vaccine (Experimental)
  Interventions: Drug: GC FLU® Injection, GC FLU® Pre-filled Syringe Injection

INTERVENTIONS:
Drug: GC FLU® Injection, GC FLU® Pre-filled Syringe Injection

SUMMARY:
This study is aimed to confirm the lot-to-lot consistency of 3 consecutive batches of 'GC FLU® Pre-filled Syringe Injection' and 'GC FLU® Injection' in the lot-to-lot

DETAILED DESCRIPTION:
This is a Post-Marketing, Multicentre, Open, Randomized Phase 4 Clinical Study. Subjects who gave voluntary written informed consent to participate in the study were screened for eligibility in the study, and those who met the eligibility criteria were randomized in the investigational group.

An investigator assessed the effectiveness (immunogenicity) and safety of the study vaccine in each subject during his/her participation in the study.

Subjects were randomized (Visit 1) into the investigational group according to a randomization table previously generated, and were vaccinated with influenza split vaccine, 'GC FLU®Pre-filled Syringe Injection' and 'GC FLU®Injection'.

12 Assessments for HI titre to each strain of influenza were performed at Visit 1 (pre-vaccination), and at Visit 3 (21 days after vaccination) for the efficacy (immunogenicity) evaluation [Picture 1].For the safety assessment, subject diaries were handed out to subjects, who were instructed to record any adverse event emerging ager the receipt of study vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults≥ 18 and < 65years of age who can be followed up for 21 days.

Depending on the part of the study that a subject was going to participate, age criteria were further divided as follows:

Lot-to-lot consistency study [PART A]: ≥ 18 to < 65 years of age Annual clinical trial [PART B]: ≥ 18 to < 65 years of age [adults]

* 65 years of age [elderly population]

  * Subjects who gave voluntary written consent to participate in the study, and are able to comply with the study requirements.

Exclusion Criteria:

* Subjects with a known hypersensitivity of allergic reaction to eggs or egg products, to chicken or chichenproducts, to any component of the study vaccine, neomycin or gentanicin.
* Subjects with immune system disorders, including immune deficiency disease.
* Subjects with a history of Guillain-Barre syndrome.
* Subjects with severe chronic disease (e.g., cardiovascular disease except for controlled hypertension, respiratory disease, metabolic disease, renal dysfunction or hemoglobinopathy, etc.) who in the investigator's opinion may have difficulty in participating in the study.
* Subjects with haemophilia or receiving a treatment with an anticoagulant, who are at increased risk of serious bleeding during intramuscular injection.
* Subjects who had acute fever with the body temperature exceeding 38.0 °C within 72 hours before vaccination with the study drug.
* Subjects who had received other vaccinations within 7 days before vaccination with the study drug, or those who had another vaccination scheduled during the study.
* Subjects who had received immunosuppressant or immune modifying drug within 3 months before vaccination with the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1139 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
GMT (Geometric Mean Titre) of HI antibody titrebefore vaccination (Day 0) and after vaccination | Day 21

SECONDARY OUTCOMES:
The percentage of subjects achieving seroconversion for HI antibody (Seroconversion rate) | Day21
GMT (Geometric Mean Titre) of HI antibody titre before vaccination (Day 0) and after vaccination | Day 21
Solicited local adverse events (topical symptoms) and solicited general adverse events (systemic symptoms) occurring from the date of vaccination until 6 days after vaccination | Day 6
The percentage of subjects achieving HI antibody titre ≥ 1:40 following the receipt of vaccination (Seroprotection rate). | Day21
The percentage of subjects achieving seroconversion for HI antibody (Seroconversion rate) | Day 21
The percentage of subjects achieving HI antibody titre ≥ 1:40 following the receipt of vaccination(Seroprotection rate). | Day 21
Unsolicited adverse events occurring from the date of vaccination until 21 days after vaccination | Day 21